CLINICAL TRIAL: NCT06628622
Title: A Phase Ib, Multi-center, Randomized, Double-blind, Parallel Group, Placebo-controlled Trial to Evaluate the Effects on Impulsivity, Pharmacokinetics, Safety, and Tolerability of Oral BI 1356225 in Patients With Opioid Use Disorder Taking Background Buprenorphine Treatment
Brief Title: A Study to Test Whether BI 1356225 Improves Impulsive Behavior in People With Opioid Use Disorder Who Are Taking Buprenorphine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1427-0015; U1111-1307-0808 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1356225 (Experimental)
  Interventions: Drug: BI 1356225
- Placebo matching BI 1356225 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356225 — BI 1356225
  Arms: BI 1356225
Drug: Placebo — Placebo
  Arms: Placebo matching BI 1356225

SUMMARY:
This study is open to people between 18 and 65 years of age with opioid use disorder. Opioid use disorder is also called opioid addiction or opioid dependence. People can join the study if they currently take a medicine called buprenorphine. People with opioid dependence can act on impulse, which can lead to risky behaviours. The purpose of this study is to find out whether a medicine called BI 1356225 improves impulse control in people with opioid dependence.

Participants are put into 2 groups by chance. One group takes BI 1356225 tablets and the other group takes placebo tablets. Placebo tablets look like BI 1356225 tablets but do not contain any medicine. Participants take a tablet once a day for 8 days. All participants also continue taking buprenorphine.

Participants are in the study for up to 6 weeks. During this time, they visit the study site 3 times. At visit 2, participants stay at the study site for 9 nights. Doctors test participants' impulsivity using tasks or games on a computer and questionnaires. The results are compared between the 2 groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, 18 to 65 years of age, both inclusively, at the time of consent
2. Meet current diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) criteria for opioid use disorder, of at least moderate severity within the 12 months prior to screening
3. Currently engaged in medications for opioid use disorder (MOUD) treatment with one of the following regimens:

   1. buprenorphine/naloxone sublingual film total daily dose ranging from 8 mg/2 mg to 24 mg/6 mg for at least 2 weeks at screening OR
   2. buprenorphine/naloxone sublingual tablet from 5.7 mg/1.4 mg to 17.1 mg/4.3 mg total daily dose for at least 2 weeks at screening OR
   3. buprenorphine sublingual tablet from 8 mg to 24 mg total daily dose for at least 2 weeks at screening OR
   4. on depot injectable buprenorphine for at least 5 weeks at screening, with at least 1 week since last depot buprenorphine injection
4. Have a current MOUD prescription in accordance with inclusion criterion 4 and a positive urine drug screen for buprenorphine during screening and upon presenting for randomization to document buprenorphine use
5. Willingness to abstain from using alcohol for 24 hours (h) and all other drugs of abuse for 72 h prior to Day 1 and through discharge from the trial site on Day 9
6. Women of child-bearing potential must be able and willing, as confirmed by the investigator, to use highly effective methods of contraception
7. Further inclusion criteria apply.

Exclusion Criteria:

1. Lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, delusional disorder, or autism spectrum disorder as confirmed by the mini international neuropsychiatric interview (MINI) at the screening visit
2. Moderate or severe substance use disorder other than opioid use disorder (OUD) within the 6 months prior to screening (excluding tobacco, caffeine, and moderate stimulant use)
3. Severe stimulant use disorder within the 3 months prior to screening
4. Any other psychiatric disorder that is not currently stable in symptoms and treatment. Stable is defined as having no significant changes in symptom acuity or treatment (medication or psychotherapy treatment) in the 8 weeks prior to randomization
5. Score of ≥20 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
6. Positive results on a urine drug screen for ≥3 drugs (not counting buprenorphine or TCAs) at screening. In the case of a positive drug screen for 1 or 2 agents, if the participant does not meet the exclusion criteria regarding substance use disorder for these compounds, they may be included if the investigator determines that use will not be an impediment to trial participation or accurate data collection
7. Any positive result on a urine drug screen (not counting buprenorphine, TCAs, or cannabis) at admission to the trial site on Day -1
8. Intoxication at screening or randomization, as determined by clinical exam and breathalyzer
9. Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-02-04 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in k parameter of the delay discounting task (DDT) on Day 8 | at baseline and at Day 8
  In the DDT, participants make choices on the screen between a smaller, immediate amount of money and a larger, delayed amount. Steep discounting of delayed rewards is indicative of cognitive impulsivity.
  The key outcome variable for this task is the discount rate (k) or rate at which delayed rewards lose their value.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Collaborative Neuroscience Research, LLC, Los Alamitos, Los Alamitos, California
  - University of California Los Angeles, Los Angeles, California
  - iResearch Atlanta, Decatur, Georgia
  - Hassman Research Institute-Marlton-66897, Marlton, New Jersey
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com